CLINICAL TRIAL: NCT02841605
Title: Enteric Nervous System in Alzheimer Disease
Acronym: ENTEROMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: RC15_0458
Record Dates: First submitted 2016-07-19; First posted 2016-07-22 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-07

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- AD group (Other): AD group: rectosigmoidospcopy with biopsies of colon
  Interventions: Procedure: Rectosigmoidoscopy with colonic biopsies
- PD group (Other): PD group: rectosigmoidospcopy with biopsies of colon
  Interventions: Procedure: Rectosigmoidoscopy with colonic biopsies
- PSP group (Other): PSP group: rectosigmoidospcopy with biopsies of colon
  Interventions: Procedure: Rectosigmoidoscopy with colonic biopsies
- Patient eligible for colorectal cancer screening (Other): Patient eligible for colorectal cancer screening: colonoscopy with biopsies of colon
  Interventions: Procedure: Colonoscopy with colonic biopsies

INTERVENTIONS:
Procedure: Rectosigmoidoscopy with colonic biopsies — Rectosigmoidoscopy with colonic biopsies performed for Alzheimer patient and both control groups Parkinson and PSP
  Arms: AD group; PD group; PSP group
Procedure: Colonoscopy with colonic biopsies — Colonoscopy with colonic biopsies performed only in patient at risk of colic cancer
  Arms: Patient eligible for colorectal cancer screening

SUMMARY:
The close homology between the central and enteric nervous systems suggests that a disease process affecting the central nervous system could also involve its enteric counterpart. The investigators have recently shown in that the enteric neurons can be readily analyzed using routine colonic biopsies. This led us to propose that the enteric nervous system could represent a unique window to assess the neuropathology in living patients with a neurodegenerative disorder. The investigators have already used this approach to show that Parkinson's disease pathology was recapitulated in a single colonic biopsy. By contrast to Parkinson's disease, the detection of Alzheimer's disease (AD) pathology in the enteric neurons has so far failed. This may be due to the low number of human tissue samples in addition to the low sensitivity of the immunohistochemical methods that were used. The aim of the current research project will be therefore to reevaluate AD pathology in a large number of human colonic samples using both a morphological and biochemical approach .

The enteric nervous system could represent a unique window to assess the neuropathology in living patients with AD. This might open the way to the development of novel AD biomarkers that will directly assess the neuropathological process.

Main Aim : To Analyze the presence of beta-amyloid pathology in the enteric nervous system (ENS) in AD patients

Secondary Aim(s):

1. To analyze and describe the presence of tau in the enteric nervous system (ENS) in AD patients
2. To assess neuronal loss in submucosal tissue in AD patients.
3. To examine Glia cells in the enteric nervous system in AD patients..

ELIGIBILITY:
Inclusion Criteria:

- AD group : Patient with early to moderate Alzheimer disease (continuum of patients with MCI due to AD and patients diagnosed with probable AD) according to NIA NAA criteria MMSE score ≥18; Has one informant or care partner; No parkinsonian syndrome No sign of lewy Body dementia

- PD group (control group 1) : Patients with Parkinson Disease according UKPDSBB criteria, No dementia sign or cognitive deficit associated to AD

- PSP group (control group 2): Patients with possible or probable Progressive supranuclear palsy group PSP according to NINDS criteria Has one informant or care partner;

- Patient eligible for colorectal cancer screening (control group 3) : No history or current neurological/degenerative condition (e.g, lewy body dementia, PD, Parkinsonian syndrome, AD…) No memory complaint with a Mac Nair score ≤15 MMSE score ≥28 ; Patient at risk of colic cancer with a colonoscopy scheduled

Exclusion Criteria:

- For all groups: History of colonic disorder (e.g inflammatory condition, adenocarcinoma) History of bleeding disorder Traitement anticoagulant ou antiagrégant en cours Treatment with anticoagulant or Platelet aggregation inhibiting drugs

- Patient with AD, PSP, PD: Any neurological/neurodegenerative condition different from the group to which it belongs (e.g other than AD for AD group or other than PD for PD group….)

- Patient eligible for colorectal cancer screening Any neurological/neurodegenerative condition (e.g lewy body dementia, Parkinsonian syndrome, PD, AD..)..

Functional colopathy or Irritable Bowel Syndrome

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2016-10; Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Presence of alpha-synuclein aggregates in colonic biopsies using immunohistochemistry | 4 months
  Alpha synuclein will be analysed by means of immunohistochemistry in colonic biopsy of patients with Alzheimer disease contrasted to patients with Parkinson disease, progressive supranuclear palsy and to patients eligible for colorectal cancer screening, as a possible biomarker of AD mirroring the cerebral anomaly.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: No